CLINICAL TRIAL: NCT04978766
Title: Early Childhood Interventions to Reduce Inequality in Educational Opportunities
Brief Title: Promoting Early Language Development Through Parent-child Book Reading in Costa Rica
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Costa Rica (Other)
Collaborators: Caja Costarricense de Seguro Social (Other Government)
Responsible Party: Principal Investigator, Ana María Carmiol, Professor of Psychology at Instituto de Investigaciones Psicológicas, Universidad de Costa Rica
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 723-B9-343; R019-SABI-00235 (Other: Ethics Committee of the Caja Costarricense del Seguro Social)
Record Dates: First submitted 2021-07-20; First posted 2021-07-27 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Language Development
Keywords: Book reading; Infancy; Interactive reading; Vocabulary development; Parenting

STUDY DESIGN:
Intervention Model Description: All participants will take baseline measures. After baseline, each participant will be randomly assigned to the control or the experimental group. At posttest, all measures taken at baseline will be evaluated again in all participants.
Who Masked: Outcomes Assessor
Masking Description: An external collaborator will create the allocation sequence for each of the two participating health centers (stratified randomization). Two independent research assistants will prepare the allocation in sequentially numbered, opaque, sealed and stapled envelopes. Aluminium foil inside each envelope will be used to render the envelope impermeable to intense light. This will allow the allocation sequence to be concealed from the researcher assessing participants at baseline. Once baseline assessment is completed, the next consecutively numbered envelope will be opened to reveal the participant's allocation.
  Treatment for the experimental group will be provided by two different researchers who will not participate in outcome assessment.
  A different researcher (outcome assessor), blind to the allocation sequence, to the participant's allocation and to the participant's baseline scores, will complete the participants' assessments during posttest.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interactive Book Reading Group (Experimental): Participants in this arm will take baseline measures, will receive the intervention and will take posttest measures.
  Interventions: Behavioral: Interactive Book Reading
- Control Group (No Intervention): Participants in this arm will take baseline and posttest measures. For ethical purposes, they will receive the intervention after posttest measures are taken.

INTERVENTIONS:
Behavioral: Interactive Book Reading — The intervention is a package including five children's books and information on how to practice interactive book reading. Information includes 36 audiovisual products delivered via text messaging over a 12-week period. Products include:
  1. An introductory video about interactive book reading, along with a written list of recommendations on how to practice interactive book reading.
  2. Two videos of child development experts explaining the benefits of interactive reading.
  3. Thirty written text messages strengthening content provided in the videos.
  4. Three audio messages guiding the progress of the intervention.
  Based on Abraham and Michie's (2008) taxonomy of behavior change techniques, one audiovisual product prompts specific goal settings, 13 provide instruction, one provides information on consequences, 10 prompt practice, three use follow-up prompts, one prompts self-monitoring of behavior, one models or demonstrates the behavior and six prompt barrier identification.
  Arms: Interactive Book Reading Group

SUMMARY:
The purpose of this study is to analyze the effect of an interactive parent-child book reading intervention. The intervention includes two components: the provision of five children's books to parent-child dyads and information about how to practice interactive book reading. The investigators expect to find an effect of this intervention on a) infants' expressive vocabulary, b) reading activity, c) parental expectations and knowledge about language development and d) parental use of interactive book reading strategies.

DETAILED DESCRIPTION:
The foundations of optimal health, growth and development are forged early in life, when income-related gaps in learning opportunities already exist in Costa Rica. It is therefore important for the government to mitigate the effects of these gaps through programs targeting the development of academic, behavioral, socioemotional and economic abilities. Key to the success of such programs is to consider physical health, nutrition, responsive care and early learning. Multiple government-led initiatives in Costa Rica had been carried out in order to provide adequate programs for infants and young children. Evidence of these efforts are observed in the low rates attained in infant mortality, malnutrition and anemia, as well as the high coverage of the current immunization program. However, policies targeting early learning in children under 36 months of age are incipient and government initiatives in this regard are relatively recent.

The purpose of this study is to promote early language development, a central component of early learning. Our goal is to implement and evaluate a low-cost intervention targeting parents of infants who benefit from the existing immunization program of the public health services offered by the Caja Costarricense del Seguro Social (Costa Rican Social Security Fund).

The investigators will use an experimental design to randomly assign 15- to 17-month-old infants and their caregivers to one of two groups: a control group or an experimental group. In the experimental group, caregivers will receive a package including five children's books and 36 text messages with information on how to practice interactive book reading with their children. This information will be delivered over a period of 12 weeks. The control group will not receive any treatment during the implementation of the intervention.

In order to measure the efficacy of the intervention, the investigators will evaluate a) infants' expressive vocabulary, b) parent-child reading activity, c) parental expectations and knowledge about language development and d) parental use of interactive book reading strategies at baseline (15-17 months of age) and at posttest (18-20 months of age) in the control and the experimental group. After posttest, the control group will receive the complete intervention.

The investigators expect to find an effect of the interactive book reading intervention on a) infants' expressive vocabulary, b) reading activity, c) parental expectations and knowledge about language development and d) parental use of interactive book reading strategies.

ELIGIBILITY:
Inclusion criteria for infants:

* Age limits: 15 months to 17 months.
* Sex: All.
* Infant was born full term (≥ 37 weeks).
* Infant is raised in a monolingual Spanish-speaking home.

Inclusion criteria for mothers:

* Mother knows how to read and write.
* Mother has access to cell phone with internet.

Exclusion Criteria:

* Neither caregivers nor infants must have any significant known physical, mental or learning disability.

Ages: 15 Months to 17 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 184 (Actual)
Dates: Start 2021-08-13 (Actual); Primary Completion 2022-09-10 (Actual); Study Completion 2022-09-10 (Actual)

PRIMARY OUTCOMES:
Change in infant expressive vocabulary | Baseline [15 to 17-months] and Posttest [18 to 20-months].
  Infant expressive vocabulary will be measured with the short form (SF) Spanish versions of the MacArthur-Bates Communicative Development Inventories (CDI). Parents will complete version I (CDI-SFI) of the inventory at baseline and version II (CDI-SFII) of the inventory at posttest. Scores on the CDI-SFI inventory range from 0 to 104. Scores on the CDI-SFII inventory range from 0 to approximately 100-135, depending on the complexity of the participant's linguistic production. For both inventories, higher scores indicate a better outcome.

SECONDARY OUTCOMES:
Change in parental report of reading activities | Baseline [15 to 17-months] and Posttest [18 to 20-months].
  Parental report of reading activities will be measured with the Spanish version of the Reading Subscale (READ) of the Cognitive Home Environment Questionnaire (StimQ-Toddler). Scores range from 0 to 19. Higher scores indicate a better outcome.
Change in parental expectations and knowledge about language development | Baseline [15 to 17-months] and Posttest [18 to 20-months].
  Parental report of expectations and knowledge about language development will be measured with the Spanish version of the Survey of Parent/Provider Expectations and Knowledge (SPEAK), a self-administered questionnaire assessing expectations and knowledge about early childhood cognitive and language development. Scores range from 0 to 54. Higher scores indicate a better outcome.
Change in parental use of interactive book reading strategies | Baseline [15 to 17-months] and Posttest [18 to 20-months].
  Video recordings of parent-child dyads reading books at baseline and posttest will be analyzed for quantity of interactive book reading strategies. Videos will be first transcribed and subsequently coded according to the following coding categories: word tokens, word types, mean length of utterance, number of questions and pointing tokens. Range of scores depends on participants' communicative/linguistic production. Higher scores indicate a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Ana M. Carmiol, PhD, Principal Investigator — Universidad de Costa Rica
Locations (2):
- Costa Rica (2):
  - Área de Salud (CCSS), Santo Domingo de Heredia, Santo Domingo, Heredia Province
  - Área de Salud (CCSS), Desamparados 2, Desamparados, Provincia de San José

IPD SHARING:
Plan to Share IPD: Yes
With participants' permission, individual participant data (IDP) will be archived in accordance with the guidelines of Costa Rican national law number 9234 (Ley de Investigación Biomédica).
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: IDP that underlies results in a publication will be shared after completion of the publication process. This process will take place in accordance with the guidelines of Costa Rican national law number 9234 (Ley de Investigación Biomédica),
Access Criteria: Under request and in accordance with the guidelines of Costa Rican law number 9234 (Ley de Investigación Biomédica).

REFERENCES:
- [Background] Jackson-Maldonado, D., Marchman, V. A., & Fernald, L. C. (2013). Short-form versions of the Spanish MacArthur-Bates Communicative Development Inventories. Applied Psycholinguistics, 34(4), 837-868.
- [Background] Mol, S. E., Bus, A. G., De Jong, M. T., & Smeets, D. J. (2008). Added value of dialogic parent-child book readings: A meta-analysis. Early education and development, 19(1), 7-26.
- [Background] Muhinyi, A., & Rowe, M. L. (2019). Shared reading with preverbal infants and later language development. Journal of Applied Developmental Psychology, 64, 101053. https://doi.org/10.1016/j.appdev.2019.101053
- [Background] Suskind, D. L., Leung, C. Y., Webber, R. J., Hundertmark, A. C., Leffel, K. R., Suskind, E., Hernandez, M. W., & Graf, E. (2018). Development of the survey of parent/provider expectations and knowledge (SPEAK). First Language, 38(3), 312-331.
- [Background] Ministerio de Salud, Instituto Nacional de Estadística y Censos, & Fondo de las Naciones Unidas para la Infancia. (2018). Encuesta de mujeres, niñez y adolescencia (EMNA).
- [Result] Abraham C, Michie S. A taxonomy of behavior change techniques used in interventions. Health Psychol. 2008 May;27(3):379-87. doi: 10.1037/0278-6133.27.3.379. PMID 18624603
- [Result] Black MM, Walker SP, Fernald LCH, Andersen CT, DiGirolamo AM, Lu C, McCoy DC, Fink G, Shawar YR, Shiffman J, Devercelli AE, Wodon QT, Vargas-Baron E, Grantham-McGregor S; Lancet Early Childhood Development Series Steering Committee. Early childhood development coming of age: science through the life course. Lancet. 2017 Jan 7;389(10064):77-90. doi: 10.1016/S0140-6736(16)31389-7. Epub 2016 Oct 4. PMID 27717614
- [Result] Cusick SE, Georgieff MK. The Role of Nutrition in Brain Development: The Golden Opportunity of the "First 1000 Days". J Pediatr. 2016 Aug;175:16-21. doi: 10.1016/j.jpeds.2016.05.013. Epub 2016 Jun 3. No abstract available. PMID 27266965
- [Result] Dreyer, B. P., Mendelsohn, A. L., & Tamis-LeMonda, C. S. (1996). Assessing the child's cognitive home environment through parental report; reliability and validity. Early Development and Parenting: An International Journal of Research and Practice, 5(4), 271-287.
- [Result] Instituto Nacional de Estadística y Censos. (2018). Mortalidad Infantil y Evolución Reciente 2018 I Semestre. Datos Preliminares. Volumen 1, Año 14.